CLINICAL TRIAL: NCT04533529
Title: A Multicenter, Double-Blind, Randomized, Parallel-Group, Placebo-Controlled, Study to Evaluate the Efficacy and Safety of Seltorexant 20 mg as Adjunctive Therapy to Antidepressants in Adult and Elderly Patients With Major Depressive Disorder With Insomnia Symptoms Who Have Responded Inadequately to Antidepressant Therapy and an Open-labeled Long-term Safety Extension Treatment With Seltorexant
Brief Title: A Study of Seltorexant as Adjunctive Therapy to Antidepressants in Adult and Elderly Participants With Major Depressive Disorder With Insomnia Symptoms Who Have Responded Inadequately to Antidepressant and Long-term Safety Extension Treatment With Seltorexant
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR108804; 2020-000337-40 (EudraCT Number); 42847922MDD3001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2020-08-14; First posted 2020-08-31 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major | interventions — seltorexant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Seltorexant (Experimental): Participants will receive seltorexant tablet orally once daily, from Day 1 to Day 42 in double blind (DB) treatment phase. Eligible participants who will enter the open label (OL) treatment phase will receive seltorexant tablet daily from OL baseline until the end of phase/ early withdrawal (EW) visit (Up to 1 Year).
  Interventions: Drug: Seltorexant
- Placebo (Placebo Comparator): Participants will receive matching placebo tablet orally once daily, from Day 1 to Day 42 in double blind (DB) treatment phase.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Seltorexant — Seltorexant tablet will be administered orally once daily.
  Other Names: JNJ-42847922
  Arms: Seltorexant
Drug: Placebo — Matching placebo tablet will be administered orally once daily.
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the efficacy of seltorexant compared with placebo as adjunctive therapy to an antidepressant in improving depressive symptoms in participants with major depressive disorder with insomnia symptoms (MDDIS) who have had an inadequate response to current antidepressant therapy with an selective serotonin reuptake inhibitor (SSRI) or serotonin-norepinephrine reuptake inhibitor (SNRI) in double-blind treatment phase and to assess the long-term safety and tolerability of seltorexant as adjunctive therapy to an antidepressant in participants with major depressive disorder (MDD) in open-label treatment phase.

DETAILED DESCRIPTION:
Major depressive disorder (MDD) is a common, serious, recurrent disorder. Seltorexant (JNJ-42847922) is a potent and selective antagonist of the human orexin-2 receptor (OX2R) that is being developed for adjunctive treatment of major depressive disorder with insomnia symptoms (MDDIS). The hypothesis for this study is that adjunctive treatment with seltorexant is superior to placebo in treating depressive symptoms, as measured by change in Montgomery Asberg Depression Rating Scale (MADRS) total score from baseline to Day 43 in adult and elderly participants with MDDIS who have had an inadequate response to treatment with a SSRI/SNRI. The study will be conducted in 4 phases: a screening phase (up to 30 days), a double-blind (DB) treatment phase (43 days), open label (OL) treatment phase (1-year), and a post treatment follow-up phase (7 to 14 days after end of treatment). The total study duration for each participant will be up to 64 weeks. Efficacy, safety, pharmacokinetics, and biomarkers will be assessed at specified time points during this study.

ELIGIBILITY:
Inclusion Criteria:

* Meet Diagnostic and Statistical Manual of Mental Disorders-5th edition (DSM-5) diagnostic criteria for major depressive disorder (MDD), without psychotic features, based upon clinical assessment and confirmed by the Structured Clinical Interview for DSM-5 Axis I Disorders-Clinical Trials Version (SCID-CT) diagnosed with first depressive episode prior to age 60. The length of the current depressive episode must be less than or equal to (<=) 24 months prior to randomization
* Have had an inadequate response to at least 1 but no more than 2 antidepressants, administered at an adequate dose and duration in the current episode of depression. The current antidepressant cannot be the first antidepressant treatment for the first lifetime episode of depression. An inadequate response is defined as less than (<) 50 percent (%) reduction but with some improvement (that is, improvement greater than [>] 0%) in depressive symptom severity with residual symptoms beyond insomnia present, and overall good tolerability, as assessed by the Massachusetts General Hospital-Antidepressant Treatment Response Questionnaire (MGH-ATRQ)
* Is receiving and tolerating well any one of the following selective serotonin reuptake inhibitor (SSRI) or serotonin-norepinephrine reuptake inhibitor (SNRI) for depressive symptoms at screening, in any formulation and available in the participating country: citalopram, duloxetine, escitalopram, fluvoxamine, fluoxetine, milnacipran, levomilnacipran, paroxetine, sertraline, venlafaxine, desvenlafaxine, vilazodone, or vortioxetine at a stable dose (at therapeutic dose level) for at least 6 weeks, and for no greater than 18 months in the current episode
* Body mass index (BMI) between 18 and 40 kilograms per meter square (kg/m^2), inclusive (BMI = weight/height^2)
* Participant must be medically stable on the basis of the following performed at screening: physical examination (including a brief neurological examination), vital signs (including blood pressure), and 12-lead electrocardiogram (ECG) performed at screening and baseline

Exclusion Criteria:

* Has a recent (last 3 months) history of, or current signs and symptoms of, a) severe renal insufficiency (creatinine clearance [CrCl] <30 milliliter per minute [mL/min]); b) clinically significant or unstable cardiovascular, respiratory, gastrointestinal, neurologic, hematologic, rheumatologic, immunologic or endocrine disorders; c) uncontrolled Type 1 or Type 2 diabetes mellitus
* Has a current or recent history of homicidal ideation or serious suicidal ideation within the past 3 months, corresponding to a positive response on item 4 (active suicidal ideation with some intent to act, without specific plan) or item 5 (active suicidal ideation with specific plan and intent) for ideation on the Columbia Suicide Severity Rating Scale (C-SSRS), or a history of suicidal behavior within the past 6 months, as validated by the C-SSRS at screening or Day 1. Participants with prior suicidal behavior in the past year, or prior serious suicidal ideation/plan within the past 6 months, should be carefully screened. For current suicidal ideation, only participants with non serious items (1-3 of the suicidal ideation section of the C-SSRS) may be included at the discretion of the investigator
* Has a history of treatment-resistant MDD, defined as a lack of response to 2 or more adequate antidepressant treatments in the current episode, as indicated by no or minimal (<25% improvement in symptoms) when treated with an antidepressant of adequate dose (per MGH-ATRQ) and duration (at least 6 weeks)
* Has history or current diagnosis of a psychotic disorder, bipolar disorder, intellectual disability, autism spectrum disorder, borderline personality disorder, or somatoform disorders
* Has any significant primary sleep disorder, including but not limited to obstructive sleep apnea, restless leg syndrome, or parasomnias. Participants with insomnia disorder are allowed
* Has a history of moderate to severe substance use disorder including alcohol use disorder according to DSM-5 criteria within 6 months before screening

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 588 (Actual)
Dates: Start 2020-09-16 (Actual); Primary Completion 2023-04-25 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Double-blind (DB) Treatment Phase: Change From Baseline in Montgomery-Asberg Depression Rating Scale (MADRS) Total Score | Baseline, Day 43
  MADRS is a clinician-administered scale designed to measure depression severity and detects changes due to antidepressant treatment. The MADRS evaluates the following 10 items: apparent sadness, reported sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, and suicidal thoughts. Each item is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), for a total possible score of 60. Higher scores represent a more severe condition.
Open-Label (OL) Treatment Phase: Number of Participants with Adverse Events (AEs) including AEs of Special Interest (AESI) as a Measure of Safety and Tolerability | 1 year
  Number of participants with AE including AE of special interest as a measure of safety and tolerability will be reported. An AE is any untoward medical occurrence in a clinical study participant administered a investigational or non-investigational medicinal product. An AE does not necessarily have a causal relationship with the treatment. AESI will comprise of cataplexy, sleep paralysis, complex, sleep-related behaviors/parasomnias, sleep terrors, bruxism, sleep sex, sleep related eating disorder, catathrenia, fall and motor vehicle accident.
OL Treatment Phase: Change From Baseline in Blood Pressure | Baseline (Day 43), up to 1 year
  Change from baseline in blood pressure will be reported.
OL Treatment Phase: Change From Baseline in Pulse Rate | Baseline (Day 43), up to 1 year
  Change from baseline in pulse rate will be reported.
OL Treatment Phase: Change From Baseline in Weight | Baseline (Day 43), up to 1 year
  Change from baseline in weight as a part of physical examination will be reported.
OL Treatment Phase: Change From Baseline in Body Mass Index (BMI) | Baseline (Day 43), up to 1 year
  Change from baseline in BMI as a part of physical examination will be reported.
OL Treatment Phase: Change From Baseline in Suicidality Assessment Using the Columbia Suicide Severity Rating Scale (C-SSRS) | Baseline (Day 43), up to 1 year
  Change from baseline in suicidality assessment using C-SSRS will be reported. C-SSRS is a clinician rated assessment of suicidal behavior and/or intent. Scale consists of 28 items in 4 sections: suicide behavior, actual attempts, suicidal ideation, and intensity of ideation. Suicidal ideation consists of 5 'yes/no' items: wish to be dead, non-specific active suicidal thoughts, active suicidal ideation with any methods (not plan) without intention to act, active suicidal ideation with some intent to act without specific plan, active suicidal ideation with specific plan and intent. Only items with yes responses are listed. Worsening of suicidal ideation indicates an increase in severity of suicidal ideation from baseline. Suicidal behavior consists of 5 'yes/no' items: preparatory acts or behavior, aborted attempt, actual attempt, completed suicide.
OL Treatment Phase: Physician Withdrawal Checklist (PWC-20) Scores | End of Treatment/Early withdrawal to end of the Follow-up visit (up to 14 days)
  Withdrawal symptoms assessment using the PWC-20 will be reported. The PWC-20 is a simple and accurate method used to assess potential withdrawal symptoms following cessation of treatment. The PWC-20 is a reliable and sensitive instrument for the assessment of discontinuation symptoms. Each individual item score ranges from 0 (not present) to 3 (severe), where higher scores = more affected condition.
OL Treatment Phase: Number of Participants with Laboratory Abnormalities | Up to 1 year
  Number of participants with laboratory abnormalities related to hematology, serum chemistry, coagulation, liver function tests and urinalysis will be reported.
OL Treatment Phase: Change From Baseline in QTc Interval | Baseline (Day 43), up to 1 year
  Change from baseline in QT interval corrected for heart rate (QTc interval) using Fridericia method will be measured by electrocardiogram (ECG).
OL Treatment Phase: Change from Baseline in Heart Rate (HR) | Baseline (Day 43), up to 1 year
  Change from baseline in HR will be measured by ECG.
OL Treatment Phase: Change from Baseline in QRS Interval | Baseline (Day 43), up to 1 year
  Change from baseline in QRS interval will be measured by ECG.
OL Treatment Phase: Change from Baseline in PR Interval | Baseline (Day 43), up to 1 year
  Change from baseline in PR interval will be measured by ECG.
OL Treatment Phase: Change From Baseline in QT Interval | Baseline (Day 43), up to 1 year
  Change from baseline in QT interval will be measured by ECG.
OL Treatment Phase: Participant-reported Sexual Functioning Using Arizona Sexual Experiences Scale (ASEX) Score | Up to 1 year
  The ASEX is a patient-reported 5-item rating scale that quantifies sex drive, arousal, vaginal lubrication/penile erection, ability to reach orgasm, and satisfaction from orgasm. The total scores range from 5 to 30, with the higher scores indicating more sexual dysfunction.

SECONDARY OUTCOMES:
DB Treatment Phase: Change From Baseline in the MADRS Without Sleep Item (MADRS-WOSI) Total Score | Baseline and Day 43
  Change from Baseline in MADRS-WOSI will be reported. MADRS-WOSI is defined as the full MADRS without the sleep item. The total score ranges from 0 to 54, with higher scores corresponding to greater symptom severity.
DB Treatment Phase: Change From Baseline in Sleep Disturbance Using the Patient Reported Outcome Measurement Information System-Sleep Disturbance (PROMIS-SD) Short Form 8a T-score | Baseline and Day 43
  The PROMIS-SD is used to assess self-reported perceptions of sleep quality, sleep depth and restoration associated with sleep. The full PROMIS-SD includes 27 items with each item based on a 7-day recall period and assessed on a 5 level Likert-type scale. The 8-item short form will be used in this study, in which responses are scored 1 to 5 for each item. A higher score on 5 of the 8 items reflects a worse outcome, whereas a higher score on 3 items reflects an improved outcome; therefore, the directionality of the 8 item scores are first synchronized prior to calculation of the total raw score. To find the total raw score for a short form with all questions answered, sum the values of the response to each question. For example, for the adult 8-item form, the lowest possible raw score is 8; the highest possible raw score is 40. Higher overall score indicates more sleep disturbance.
DB Treatment Phase: Change From Baseline in the MADRS-6 Total Score | Baseline and Day 43
  The MADRS-6 scale is a clinician-administered questionnaire used to measure the severity of MDD symptoms. The MADRS-6 scale is a subset of the MADRS-10 scale, comprises of the following individual questionnaire items: Apparent Sadness, Reported Sadness, Inner Tension, Lassitude, Inability to Feel, and Pessimistic Thoughts. Scores range from 0 (no apparent symptoms) to 36 (most severe symptoms).
DB Treatment Phase: Percentage of Participants with Response on Depressive Symptoms Scale Based on Montgomery-Asberg Depression Rating Scale (MADRS) | Day 43
  Percentage of participants with response on depressive symptoms scale based on MADRS will be reported. Responders are defined as percentage of participants with greater than or equal to (>=) 50 percent (%) improvement in the MADRS total score from baseline to Day 43.
DB Treatment Phase: Change From Baseline in Patient Health Questionnaire, 9-Item (PHQ-9) Total Score | Baseline and Day 43
  The PHQ-9 is a 9-item, participant reported outcome measure to assess depressive symptoms. The scale scores each of the 9 symptom domains of the diagnostic and statistical manual of mental disorders-5th edition (DSM-5) major depressive disorder (MDD) criteria. Each item is rated on a 4 point scale (0=not at all, 1=several days, 2=more than half the days, and 3=nearly every day). The participant's item responses are summed to provide a total score (range of 0 to 27), with higher scores indicating greater severity of depressive symptoms.
DB Treatment Phase: Number of Participants with Adverse Events (AEs) including AEs of Special Interest (AESI) as a Measure of Safety and Tolerability | Up to Day 50 to 57 (every two weeks)
  Number of participants with AE including AE of special interest as a measure of safety and tolerability will be reported. An AE is any untoward medical occurrence in a clinical study participant administered a investigational or non-investigational medicinal product. An AE does not necessarily have a causal relationship with the treatment. AESI include: Cataplexy, Sleep paralysis, complex, sleep-related behaviors/parasomnias such as: confusional arousal, somnambulism, sleep terror, bruxism, sleep sex, sleep-related eating disorder, sleep behavior disorder, catathrenia.
OL Treatment Phase: Change From Baseline Over Time in Montgomery-Asberg Depression Rating Scale (MADRS) Total Score | Baseline (Day 43), up to 1 year
  MADRS is a clinician-administered scale designed to measure depression severity and detects changes due to antidepressant treatment. The MADRS evaluates the following 10 items: apparent sadness, reported sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, and suicidal thoughts. Each item is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), for a total possible score of 60. Higher scores represent a more severe condition.
OL Treatment Phase: Change From Baseline Over Time in the Clinical Global Impression-Severity (CGI S) Score | Baseline (Day 43), up to 1 year
  The CGI-S is a 7-point global assessment scale that measures the clinician's impression of the severity of illness exhibited by a participant, rating according to: 1=normal (not at all ill); 2=borderline ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; and 7=among the most extremely ill participants. Higher scores indicate worsening.
OL Treatment Phase: Change from Baseline Over Time in the MADRS-WOSI Total Score | Baseline (of OL phase), up to 1 year
  Change from Baseline in MADRS-WOSI will be reported. MADRS-WOSI is defined as the full MADRS without the sleep item. The total score ranges from 0 to 54, with higher scores corresponding to greater symptom severity.
OL Treatment Phase: Change From Baseline Over Time in Sleep Disturbance Using the PROMIS SD Short Form 8a T-score | Baseline (Day 43), up to Year 1
  The PROMIS-Sleep Disturbance (PROMIS-SD) is used to assess self-reported perceptions of sleep quality, sleep depth and restoration associated with sleep. The full PROMIS-SD includes 27 items with each item based on a 7-day recall period and assessed on a 5 level Likert-type scale. The 8-item short form will be used in this study, in which responses are scored 1 to 5 for each item. A higher score on 5 of the 8 items reflects a worse outcome, whereas a higher score on 3 items reflects an improved outcome; therefore, the directionality of the 8 item scores are first synchronized prior to calculation of the total raw score. To find the total raw score for a short form with all questions answered, sum the values of the response to each question. For example, for the adult 8-item form, the lowest possible raw score is 8; the highest possible raw score is 40. Higher overall score indicates more sleep disturbance.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (122):
- United States (51):
  - Advanced Research Center Inc, Anaheim, California
  - Synexus, Cerritos, California
  - Irvine Clinical Research, Irvine, California
  - Omega Clinical Trials LLC, La Habra, California
  - Synergy East, Lemon Grove, California
  - Semel Institute for Neuroscience and Human Behavior, Los Angeles, California
  - Catalina Research Institute, Montclair, California
  - Pacific Research Partners, Oakland, California
  - North County Clinical Research, Oceanside, California
  - Syrentis Clinical Research, Santa Ana, California
  - Viking Pharmaceutical Trials Inc. dba Viking Clinical Research, Temecula, California
  - Connecticut Clinical Trials LLC, Cromwell, Connecticut
  - University of Connecticut Health Center, Farmington, Connecticut
  - Sarkis Clinical Trials, Gainesville, Florida
  - Clinical NeuroScience Solutions Inc, Jacksonville, Florida
  - Pharmax Research Clinic Inc, Miami, Florida
  - Medical Research Center of Miami II Inc, Miami, Florida
  - Phoenix Medical Research, Inc., Miami, Florida
  - Galiz Research, Miami Springs, Florida
  - Bravo Health Care Center, North Bay Village, Florida
  - APG Research LLC, Orlando, Florida
  - Combined Research Orlando, Orlando, Florida
  - Nova Psychiatry INC, Orlando, Florida
  - Revive Research Institute, Elgin, Illinois
  - Joliet Center for Clinical Research, Joliet, Illinois
  - Baber Research Group, Naperville, Illinois
  - American Medical Research, Inc., Oak Brook, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Louisiana Clinical Research, Shreveport, Louisiana
  - Adams Clinical, Watertown, Massachusetts
  - Neurobehavioral Medicine Group, Bloomfield Hills, Michigan
  - Midwest Research Group - St. Charles Psychiatric Associates, Saint Charles, Missouri
  - Mid-America Clinical Research, LLC, St Louis, Missouri
  - PsychCare Consultants Research, St Louis, Missouri
  - Premier Psychiatric Research Institute, LLC, Lincoln, Nebraska
  - Altea Research Institute, Las Vegas, Nevada
  - Hassman Research Institute, LLC., Berlin, New Jersey
  - Synexus Clinical Research US Inc, Jamaica, New York
  - Bioscience Research LLC, Mount Kisco, New York
  - Haidar Almhana Nieding, Avon Lake, Ohio
  - The Ohio State University, Columbus, Ohio
  - Lindner Center of Hope, Mason, Ohio
  - Oklahoma Clinical Research Center, Oklahoma City, Oklahoma
  - Lehigh Center for Clinical Research, Allentown, Pennsylvania
  - University of Pennsylvania - Perelman School of Medicine, Philadelphia, Pennsylvania
  - Relaro Medical Trials, Dallas, Texas
  - North Texas Clinical Trials, Fort Worth, Texas
  - Baylor College of Medicine, Houston, Texas
  - Red Oak Psychiatry Associates, Houston, Texas
  - Alpine Research Organization, Clinton, Utah
  - Green Mountain Research Institute, Rutland, Vermont
- Brazil (8):
  - CPN - Centro de Pesquisa em Neurociências Ltda, Belo Horizonte
  - CCB Centro Cardiologico de Brasilia Ltda - CCB Cardiologia, Brasília
  - Instituto de Neurologia de Curitiba, Curitiba
  - Universidade Federal do Ceara Hospital Universitario Walter Cantidio, Fortaleza
  - Instituto Mederi de Pesquisa e Saude, Passo Fundo
  - Ruschel Medicina e Pesquisa Clínica Ltda, Rio de Janeiro
  - SPDM - Associacao Paulista para o Desenvolvimento da Medicina - Hospital Sao Paulo, São Paulo
  - Instituto Bairral de Psiquiatria, São Paulo
- Bulgaria (11):
  - Mental Health Center Prof. Dr. Ivan Temkov, Burgas
  - Ambulatory for Individual Practice for Specialized Medical Care in Psychiatry Dr. Ivo Natsov ET, Cherven Bryag
  - State Psychiatric Hospital Kardzhali, Kardzhali
  - Medical center Spectar - Plovdiv EOOD, Plovdiv
  - UMHAT 'Sv. Georgi' EAD, Plovdiv
  - MHC - Sofia, EOOD, Slivnitsa
  - Medical Center St. Naum, Sofia
  - DCC 'Sv. Vrach and Sv. Sv. Kuzma and Damyan', OOD, Sofia
  - Medical Center Intermedica, OOD, Sofia
  - Medical center - VAS OOD, Targovishte
  - Mental Health Center - Vratsa EOOD, Vratsa
- Colombia (5):
  - Centro de Investigaciones y Proyectos en Neurociencias CIPNA, Barranquilla
  - HOMO - ESE Hospital Mental de Antioquia, Bello
  - Centro de Investigaciones del Sistema Nervioso Grupo Cisne Ltda., Bogotá
  - Fundacion Centro de Investigacion Clinica CIC, Medellín
  - Psynapsis Salud Mental S.A., Pereira
- Czechia (5):
  - BRAIN-SOULTHERAPY s.r.o., Kladno
  - Neuroterapie KH S R O, Kutná Hora
  - A Shine S R O, Pilsen
  - Clintrial s r o, Prague
  - Medical Services Prague S R O, Prague
- Mexico (3):
  - Iecsi S.C., Monterrey
  - CRI Centro Regiomontano de Investigacion SC, Nuevo León
  - Bind Investigaciones S.C., San Luis Potosí City
- Russia (8):
  - Psychoneurological Dispensary of Frunzensky District, Saint Petersburg
  - SPb SBIH 'City Psychoneurological Dispensary # 7 (With Inpatient Facilities)', Saint Petersburg
  - City Psychiatric Hospital of St. Nikolay Chudotvorets, Saint Petersburg
  - Bekhterev Psychoneurological Research Institute, Saint Petersburg
  - St-Petersburg Bekhterev Psychoneurological Research Institute, Saint Petersburg
  - Psychoneurological dispensary 1, Saint Petersburg
  - Stavropol Region Psychiatric Hospital #2, Stavropol
  - Yaroslavl Region Clinical Psychiatric Hospital, Yaroslavl
- South Africa (8):
  - Farmovs Pty Ltd, Bloemfontein
  - Iatros International, Bloemfontein
  - Cape Town Clinical Research Centre, Cape Town
  - Flexivest 14 Research, Cape Town
  - DJW Research, Krugersdorp
  - Stanza Clinical Research Centre : Mamelodi, Mamelodi East
  - Synexus Watermeyer, Pretoria
  - Somerset West Clinical Research Unit, Strand
- Spain (10):
  - Institucion Hosp Hestia Palau, Barcelona
  - Hosp Univ Vall D Hebron, Barcelona
  - Hosp. Univ. de Basurto, Bilbao
  - Hosp. Univ. Ramon Y Cajal, Madrid
  - Hosp. Univ. La Paz, Madrid
  - Centro Salud Mental La Corredoria, Oviedo
  - Clinica Univ. de Navarra, Pamplona
  - Corporacio Sanitari Parc Tauli, Sabadell
  - Centro de salud San Juan - IBSAL, Salamanca
  - Hosp. Prov. de Zamora, Zamora
- Sweden (6):
  - Affecta Pskyiatrimottagning, Halmstad
  - PharmaSite Helsingborg, Helsingborg
  - ProbarE i Lund AB, Lund
  - PharmaSite, Malmo
  - Läkarmottagningen, Skövde
  - ProbarE i Solna, Stockholm
- Taiwan (7):
  - Chang-Gung Memorial Hospital-Keelung, Keelung
  - National Taiwan University Hospital, Taipei
  - Mackay Memorial Hospital, Taipei
  - Taipei Medical University, Taipei
  - Cheng Hsin General Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital- Linkou, Taoyuan

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency